CLINICAL TRIAL: NCT00513058
Title: Phase I Study Evaluating the Combination of Lapatinib + Vinorelbine in Patients With Locally Advanced or Metastatic Breast Cancer Overexpressing HER2
Brief Title: Lapatinib and Vinorelbine in Treating Women With HER2-Overexpressing Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558406; FRE-FNCLCC-GEP-01/0506 (Other: UNICANCER); 2005-005167-28 (EudraCT Number)
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lapatinib + vinorelbine (Experimental): * starting with loading dose of lapatinib per os for 7 days
  * then, combining lapatinib (oral daily continuous) + vinorelbine (intravenous, day 1 and 8 every 3 weeks)
  Interventions: Drug: Lapatinib; Drug: vinorelbine

INTERVENTIONS:
Drug: Lapatinib — Dose level (DL) 1 : 750 mg/d DL2, DL3, DL4: 1000 mg/d DL5, DL7, DL8: 1250 mg/d DL6: 1500 mg/d
  Other Names: TYVERB
Drug: vinorelbine — DL1, DL2: 20 mg/m2 DL3: 22.5 mg/m2 DL4, DL5, DL6: 25 mg/m2 DL7: 27.5 mg/m2 DL8: 30 mg/m2
  Other Names: NAVELBINE

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with vinorelbine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib and vinorelbine in treating women with HER2-overexpressing locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tolerability and feasibility of the lapatinib ditosylate and vinorelbine ditartrate combination by determining the maximum tolerated dose of vinorelbine ditartrate in combination with a biologically active dose of lapatinib ditosylate.

Secondary

* Determine the maximum administered dose.
* Investigate the pharmacokinetic interactions related to the combination of vinorelbine ditartrate and lapatinib ditosylate.
* Determine the toxicity of vinorelbine ditartrate and lapatinib ditosylate.
* Determine the objective response rate in patients with measurable lesions.
* Validate the safety and efficacy of the oral vinorelbine ditartrate and lapatinib ditosylate combination, according to the vinorelbine ditartrate oral/IV dose equivalence.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral lapatinib ditosylate on days -7 to 21 for course 1 and on days 1-21 for all other courses. Patients also receive vinorelbine ditartrate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-9 patients receive escalating doses of lapatinib ditosylate and vinorelbine ditartrate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 9 patients experience dose-limiting toxicity during course 1.

Once the MTD is determined for oral lapatinib ditosylate and IV vinorelbine ditartrate, an additional cohort of 9 patients receive oral vinorelbine ditartrate with oral lapatinib ditosylate as above.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced breast cancer (metastatic or locally advanced)
* Tumor overexpressing HER2 (HER2 3+ by IHC OR HER2 2+ by IHC and FISH positive) in samples from the primary and/or secondary tumor
* Measurable or evaluable disease
* Cancer is progressive after treatment with at least 1 line or, at most, 2 lines, of chemotherapy that included trastuzumab (Herceptin®)
* Patients presenting with treated asymptomatic cerebral metastases or leptomeningeal metastases may be included if they are neurologically stable and have not received steroids or anticonvulsant treatment for at least 4 weeks before study entry

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Female
* Menopausal status not specified
* Patients must have an estimated survival of at least 3 months
* WHO performance status (ECOG) 0-2
* Hemoglobin ≥ 9 g/dL
* ANC ≥ 1,500/mm³
* Platelets ≥ 100,000/mm³
* Total bilirubin ≤ 2.5 mg/dL
* ALT and AST ≤ 3 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 40 mL/min
* LVEF ≥ 50% (echographic or isotopic method)
* Potentially reproductive patients must agree to use an effective contraceptive method while on study treatment
* Patients must be affiliated with a Social Security system

Exclusion criteria:

* Uncontrolled cardiac pathology
* Dysphagia or inability to swallow the vinorelbine ditartrate soft capsules
* Malabsorption syndrome or disease significantly affecting gastrointestinal function
* Preexisting neuropathy (grade ≥ 2)
* Pregnant women, women who are likely to become pregnant, or women who are breastfeeding
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Individuals deprived of liberty

Exclusion criteria:

* Prior major resection of stomach or proximal bowel that could affect absorption of oral drugs
* Prior vinorelbine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | during the first cycle of treatment

SECONDARY OUTCOMES:
Pharmacokinetic interactions between vinorelbine ditartrate (oral or IV) and lapatinib ditosylate | during the first cycle of treatment
Tumor response as assessed by RECIST criteria after every 2 courses | during 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (5):
- France (5):
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Curie Hopital, Paris
  - Centre Rene Huguenin, Saint-Cloud
  - Institut Claudius Regaud, Toulouse